CLINICAL TRIAL: NCT03144271
Title: A Randomised, Double-blind, Placebo-controlled, Dose Escalation Trial of Single Subcutaneous Doses of NNC 0113-0217 to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics in Healthy Male Subjects
Brief Title: Dose Escalation Trial of Single Subcutaneous Doses of NNC 0113-0217 to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-1820; 2007-000303-15 (EudraCT Number); U1111-1193-6996 (Other: World Health Organization (WHO))
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NNC 0113-0217 (Experimental): Dose-escalation trial
  Interventions: Drug: semaglutide
- Placebo (Placebo Comparator): Dose-escalation trial
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: semaglutide — A single dose of 0.625, 1.25, 2.5, 5, 10, 20, 40 or 80 μg/kg semaglutide will be administered subcutaneously (s.c. under the skin).
  Other Names: NNC 0113-0217
  Arms: NNC 0113-0217
Drug: Placebo — A single dose of placebo will be administered subcutaneously (s.c. under the skin)
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to assess the safety and tolerability of ascending single s.c. doses of NNC 0113-0217 in healthy male subjects, aiming at establishing the Maximum Tolerated Dose (MTD)

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject)
* Subject is male
* Age 18-65 years, both included
* Body Mass Index (BMI) below 35.0 kg/m^2 (Body weight between 50 kg -150 kg, both inclusive)
* Good general health based on medical history, physical examination including ECG (Electrocardiogram) and laboratory analysis, as judged by the investigator

Exclusion Criteria:

* Previous participation, defined as randomised, in any other clinical trial involving this or other investigational products within the last 3 months before dosing
* Patients with MI (Myocardia-Infarction) during the last 12 month
* Patients receiving ACE (Angiotensin-Converting Enzyme) inhibitors, beta-blockers, thiazide diuretics, thyroid hormones, and/or lipid lowering medication who are not on a stable dose for more than 6 weeks prior to start of the study
* Use of weight lowering medications (orlistat, sibutramine, rimonabant, phentermine)
* Clinically significant GI (Gastro-Intestinal) disease including inflammatory bowel disease, irritable bowel syndrome, celiac disease, dyspepsia, apparent diabetic gastro paresis, diabetic diarrhoea, or surgery of the gastro-intestinal tract (except appendectomy and cholecystectomy)
* Subjects who are sexually active and have not been surgically sterilised must be informed that they and their partner use a highly effective method of contraception (Pearl Index below 1%) such as implants, injectables, combined oral contraceptives, or hormonal IUDs (intrauterine devices), or refrain from sexual intercourse during the study and until 1 month after completion of the trial. This is to prevent the possibility of a pregnancy from spermatocytes that can potentially be damaged by study medication
* Current treatment with drugs known to interfere with glucose metabolism such as systemic corticosteroids, non-selective beta-blockers, and MAO (Mono-Amino-Oxidase) inhibitors
* Subjects who drink more than 8 cups of tea/coffee per day
* History of drug or alcohol abuse (defined as intake of more than 28 units weekly - 1 unit = 12 oz or 360 ml of beer; 5 oz ir 150 ml of wine; 1.5 oz or 45 ml of distilled spirits)
* Alcohol intake within 48 hours prior to dosing
* Evidence of drug abuse on urine testing and serum at study entry
* The subject smokes 7 cigarettes or more, or the equivalent, per day and is unable to refrain from smoking during 3 days prior to the dosing day and during the confinement period
* Hepatitis B surface antigen (HBsAg), Hepatitis C antibodies or HIV-positive
* Impaired hepatic function measured as ALAT (Alanine aminotransferase), ASAT (Aspartate aminotransferase), alkaline phosphatase above three times the upper reference limit (one retest within one week is permitted, the last result being conclusive)
* Clinical significant abnormal laboratory test results during the screening as judged by the Investigator
* Impaired renal function, defined as s-creatinine above or equal to 135 μmol/L (=1.5mg/dL) (one retest within one week is permitted, the last result being conclusive)
* Cardiac problems defined as: decompensated heart failure (NYHA (New York Heart Association) class III and IV) at any time and/or angina pectoris and/or myocardial infarction within the last 12 months
* Blood pressure in supine position at the screening examination above 160 mmHg systolic or 90 mmHg diastolic or heart rate outside the range of 50 - 90 bpm
* Known or suspected allergy to trial product or related products
* History of significant drug allergy or drug hypersensitivity
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Blood donation or considerable blood loss - more than 500 mL, during the 3 months prior to study start
* Any condition that the investigator and / or sponsor feels would interfere with study participation or evaluation of results
* Use of non-prescription drugs, except routine vitamins, within 1 week prior to the dose of the test drug. Occasional use of paracetamol is permitted
* Subjects who have taken part in strenuous exercise within 4 days prior to trial start, due to interference with the hepatic microsomal mono-oxygenase system. The evaluation whether strenuous exercise has been undertaken will be evaluated by the Investigator, and strenuous exercise is not allowed during the trial

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-06-11 (Actual); Primary Completion 2007-10-08 (Actual); Study Completion 2007-10-08 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | After 24-33 days

SECONDARY OUTCOMES:
Area under the curve of NNC 0113-0217 | From 0-48 hours after dosing
Area under the curve of NNC 0113-0217 | From 0-168 hours after dosing
Morning fasting plasma glucose | At visit 1 (days -28 to -1), 2 (days 0-8), 3 (days 11-13) and 4 (days 17-19)
Morning fasting insulin | At visit 1 (days -28 to -1), 2 (days 0-8), 3 (days 11-13) and 4 (days 17-19)
Morning fasting glucagon | At visit 1 (days -28 to -1), 2 (days 0-8), 3 (days 11-13) and 4 (days 17-19)

CONTACTS AND LOCATIONS:
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com